CLINICAL TRIAL: NCT02571790
Title: Virtual Reality and Relaxation for the Treatment of Generalized Anxiety Disorders: a Comparative Study With Standard Relaxation
Acronym: Relax-TAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-23
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Generalized Anxiety Disorders
Keywords: Patient with Generalized Anxiety Disorders
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relaxation optimized virtual reality (Experimental): six relaxation sessions with virtual reality
  Interventions: Behavioral: Relaxation optimized virtual reality
- Classical relaxation (without Virtual Reality). (Experimental): six relaxation sessions without virtual reality
  Interventions: Behavioral: Classical relaxation (without Virtual Reality)

INTERVENTIONS:
Behavioral: Relaxation optimized virtual reality
  Arms: Relaxation optimized virtual reality
Behavioral: Classical relaxation (without Virtual Reality)
  Arms: Classical relaxation (without Virtual Reality).

SUMMARY:
The purpose is threefold: Assess the anxiety reduction, the mood positive effect and the rise of quality of life when using methods of relaxation combined with virtual reality with patients suffering from generalized anxiety disorder in comparison of the effect of traditional relaxation therapy. Observe and evaluate the effect of perceived presence in synthetic environments in the virtual experience of relaxation. Evaluate the therapeutic efficacy of stereoscopy during exposure to relaxing virtual environments for the treatment of generalized anxiety disorder.

It is a comparative, randomized, two groups study (29 in each group):

* Relaxation optimized virtual reality
* Classical relaxation (without Virtual Reality). The protocol comprised for each groups 7 relaxing sessions (with or without virtual reality epending on the group). Each session lasted for approximately 30 to 35 minutes, including a 5-minute pause between immersive trials, in order to avoid cyber sickness in the virtual reality group.

Expected results: a measurable therapeutic improvement produced by the combination of relaxation and virtual and its additional effect when compared to the traditional treatment.

Measurements of variables and therapeutic effects will be carried out with psychometric measures.

The creation process of the relaxing virtual environments has already been completed. The virtual environments are ready for use.

The apparatus needed and in our possession include:

* A laptop for generating virtual environments
* A stereoscopic display
* Apparatus for physiological measurements

ELIGIBILITY:
Inclusion Criteria:

* Male or Female.
* Age 18-65 years inclusive.
* Generalized Anxiety Disorders primary diagnosis in patients according with major depressive episode V (DSM-V) criteria.
* Topic speaking English or French language
* Subject who have signed a written informed consent and undertaking to comply with the instructions of the protocol.

Exclusion Criteria:

* Subject not having at least one inclusion criterion;
* Minor Subject, pregnant or nursing women, about not being affiliated to the social security scheme, or deprived of liberty subject;
* Age greater than 18 and less than 65 years.
* Subject Trust;
* Subject indication against having a virtual reality: epilepsy, major organ failure, severe myopia, acute psychiatric disorder (such as schizophrenia in acute period, paranoia, manic, or melancholic major depression).
* Subject did not sign the informed consent, or topic for which the legal representative has not signed this consent in cases where the subject is under curatorship.
* Subject wishing to interrupt his participation in the study before the end;
* Subject for which the occurrence of an event makes it necessary to interrupt the therapy program before the end
* History of neurological disease, head injury or mental retardation.
* Presence of a psychotic disorder decompensated
* Presence of addictologique comorbidity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
scores on psychometric scales in connection with the Generalized Anxiety Disorders (TAG) | 24 months
  Penn State Worry Questionnaire

SECONDARY OUTCOMES:
Short self-completion questionnaire on the Generalized Anxiety Disorders (TAG) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France